CLINICAL TRIAL: NCT06856629
Title: The Immediate Physiological and Perceptual Response to Blood-flow Restricted Strength Training With Eccentric Loading (E-BFR): a Randomised Crossover Study in Healthy Subjects
Brief Title: The Immediate Physiological and Perceptual Response to Blood-flow Restricted Strength Training With Eccentric Loading
Acronym: E-BFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dario Kohlbrenner (Other)
Responsible Party: Sponsor-Investigator, Dario Kohlbrenner, Principal Investigator, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BASEC2024-02223; SNCTP000006261 (Other: kofam)
Record Dates: First submitted 2025-02-06; First posted 2025-03-04 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: Blood-flow restriction training; acute physiological response; eccentric training

STUDY DESIGN:
Intervention Model Description: With random sequence allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eccentric blood-flow restriction trainig (Experimental)
  Interventions: Other: Eccentric blood-flow restriction training
- Eccentric free-flow training (Active Comparator)
  Interventions: Other: Eccentric free-flow training

INTERVENTIONS:
Other: Eccentric blood-flow restriction training — Eccentric blood-flow restriction training
  Arms: Eccentric blood-flow restriction trainig
Other: Eccentric free-flow training — Eccentric free-flow training
  Arms: Eccentric free-flow training

SUMMARY:
Decreasing workloads in strength training makes it more tolerable for a broad range of people. When designed as blood-flow restriction training, similar gains in strength and muscle mass are achieved compared to traditional training. Adding high training loads to blood-flow restriction training only in the eccentric phase (BFR-ECC) might achieve superior gains in muscle strength while still maximizing tolerability of the training stimuli.

This study aims to investigate the acute physiological and perceptual response of blood-flow restriction training with eccentric loading in comparison to traditional eccentric training. The study recruits healthy individuals ≥ 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Clinically Healthy

Exclusion Criteria:

* Physical or intellectual impairment precluding informed consent or protocol adherence
* Pain during exercise of any origin
* History of thromboembolic event in the lower extremity
* Known pregnancy (no testing is carried out)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
minute ventilation | During the intervention (i.e., exercise) for 10 minutes
  recorded with breath-by-breath analysis

SECONDARY OUTCOMES:
Other variables from breath-by-breath analysis | During the intervention (i.e., exercise) for 10 minutes
  VO2, VCO2, RER, breath rate, heart rate
Rate of perceived exertion | Immediately after the intervention (i.e., exercise)
  Numeric rating scale from 0-10. Participants rate perceived leg exertion and perceived respiratory exertion
Near-infrared spectroscopy of the vastus lateralis | During the intervention (i.e., exercise) for 10 minutes
  Tissue saturation
Delayed onset muscle soreness | 24, 48, and 72 hours after each of the intervention (i.e., exercise)
  Numeric rating scale 0-10 rating intensity of DOMS symptoms
Feasibility and tolerability | After study completion (i.e., after the second study visit, up to 2 weeks)
  Custom-made questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request